CLINICAL TRIAL: NCT02497053
Title: Four Versus Six Cycles of Pemetrexed/Platinum as a First Line Treatment of Malignant Pleural Mesothelioma; a Randomized Phase II Study
Brief Title: Four Versus Six Cycles of Pemetrexed/Platinum for MPM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omar Abdel-Rahman, Lecturer of clinical Oncology, Faculty of medicine, Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Meso-01
Record Dates: First submitted 2015-07-10; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: MPM
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Four cycles of pemetrexed/platinum
  Interventions: Drug: pemetrexed/platinum chemotherapy
- Arm B (Active Comparator): Six cycles of pemetrexed/platinum
  Interventions: Drug: Pemetrexed/platinum chemotherapy

INTERVENTIONS:
Drug: pemetrexed/platinum chemotherapy — Four cycles of pemetrexed/platinum chemotherapy
  Arms: Arm A
Drug: Pemetrexed/platinum chemotherapy — Six cycles of pemetrexed/platinum chemotherapy
  Arms: Arm B

SUMMARY:
The prognosis of mesothelioma is generally poor. The median survival of patients with unresectable malignant mesothelioma ranges approximately between 6-12 months. Survival is poor because there is no curative treatment.

Treatment options include surgery, chemotherapy and radiotherapy. Recently multimodality treatment regimens have been reported to prolong survival. Other new therapeutic approaches include immunotherapy, gene therapy, hyperthermic chemoperfusion of the pleura and photodynamic therapy, but the results have not yet been completely validated. Even with the introduction of this new therapeutic protocol, the response does not exceed 41%, with a mean survival of 12 months. The current standard of care for unresectable malignant pleural mesothelioma is pemetrexed/cisplatin. This regimen was compared to cisplatin alone in a study including 448 patients from 19 countries which was the largest trial to date among patients suffering from malignant mesothelioma. Results showed statistically significant increase in overall survival by about 30 % (12.1 months for pemetrexed /cisplatin versus 9.3 months for cisplatin alone. In addition, there was an improvement in lung function (forced vital capacity) in the pemetrexed /cisplatin arm in comparison to the cisplatin arm.

Until now, however, there is no consensus on the number of cycles of pemetrexed/cisplatin in malignant mesothelioma and there are no approved predictive markers for response.

Pemetrexed/cisplatin regimen is an expensive regimen and associated with considerable toxicity and so we need to rationalize its use in our Egyptian patients.

Therefore, the investigators aim in this work to compare 4 cycles versus 6 cycles of pemetrexed/cisplatin in malignant mesothelioma and to identify a predictive marker for response.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of malignant pleural Mesothelioma
2. No prior chemotherapy.
3. ECOG less than or equal to 2 .
4. Measurable disease according to the requirements of SWOG criteria.
5. Age ≥ 18 years .
6. Estimated life expectancy of at least 12 weeks .
7. Adequate bone marrow reserve (white blood cells [WBC] ≥ 3.5 × 109 /L, neutrophils ≥ 1.5 × 109 /L, platelets ≥ 100 × 109 /L, and hemoglobin ≥ 9.0 gm/dL).

Exclusion Criteria:

1. Presence of central nervous system metastases.
2. Inadequate liver function (bilirubin > 1.5 times upper normal limit [UNL] and alanine transaminase [ALT] or aspartate transaminase [AST] > 3.0 UNL or up to 5.0 UNL in the presence of hepatic metastases).
3. Inadequate renal function (creatinine > 1.25 times UNL, creatinine clearance < 50mL/min).
4. Serious concomitant systemic disorder incompatible with the study.
5. Second primary malignancy (except in situ carcinoma of the cervix, adequately treated basal cell carcinoma of the skin, T1 vocal cord cancer in remission, or prior malignancy treated more than 5 years prior to enrollment without recurrence).
6. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | one year

SECONDARY OUTCOMES:
Overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Omar Abdel-Rahman, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt